CLINICAL TRIAL: NCT06648473
Title: Repeatability of Magnetic Resonance Imaging in Patients With IDH1 Mutant Glioma on Ivosidenib
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor withdrew funding
Sponsor: Duke University (Other)
Collaborators: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO00116521
Record Dates: First submitted 2024-10-11; First posted 2024-10-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Low Grade Glioma of Brain
Keywords: IDH1 Mutant; ivosidenib; Pro00116521; low grade glioma; MRI
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Magnetic Resonance Imaging (MRI) Scan (Experimental): Subjects will begin the MRI with T1-pre, T2w, and volumetric 3D Fluid Attenuated Inversion Recovery (FLAIR) images being obtained. The subject will be brought out of the MRI magnet and moved into a seated position and will then have a standard Brain Tumor Imaging Protocol MRI scan.
  Interventions: Diagnostic Test: MRI Scan

INTERVENTIONS:
Diagnostic Test: MRI Scan — Subjects will begin the MRI with T1-pre, T2w, and volumetric 3D FLAIR images being obtained. The subject will be brought out of the MRI magnet and moved into a seated position and will then have a standard Brain Tumor Imaging Protocol MRI scan.

SUMMARY:
The purpose of this study is to evaluate the repeatability of magnetic resonance imaging (MRI) in patients with isocitrate dehydrogenase 1 (IDH1) mutant (mIDH1) low-grade diffuse glioma [World Health Organization (WHO) grade 2] who are receiving off-label ivosidenib.

DETAILED DESCRIPTION:
40 adult patients with histologically low-grade mIDH1 glioma (WHO grade 2) who are being seen at Duke Preston Robert Tisch Brain Tumor Center (PRTBTC) for treatment or evaluations, will be included in this protocol. Patients included in this protocol must currently be receiving off-label ivosidenib per recommendation of their treating physician and must be scheduled to receive a routine contrast-enhanced brain Magnetic Resonance Imaging (MRI) scan as part of their clinical care. The images from the routine MRI scan will be obtained as part of the patient's clinical care and will only be used in this research study if the patient agrees to be on-study by signing the informed consent form (ICF).

Subjects will undergo a routine Brain Tumor Imaging Protocol MRI scan with additional imaging sequences, in order to create a database of short interval "coffee break" repeat MRI sets. Subjects will begin their MRI by having T1-pre, T2w, and volumetric 3D Fluid Attenuated Inversion Recovery (FLAIR) images. The subject will be brought out of the magnet, sat up and then have the standard Brain Tumor Imaging Protocol MRI scan performed.

Subjects will remain on this study for the one day during which they are scheduled to receive their MRI scan

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures
2. Scheduled for contrast-enhanced magnetic resonance imaging (MRI) as part of clinical care
3. Histologically IDH1 mutant low-grade glioma (WHO grade 2) and actively receiving ivosidenib
4. Active patient treatment or evaluations at the Preston Robert Tisch Brain Tumor Center at Duke
5. Age ≥18 years and ≤70 years
6. Karnofsky performance index ≥70%
7. Primary treating physician approval

Exclusion Criteria:

1. Inability to have MRIs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Repeatability | 1 year
  Bland-Altman repeatability will be measured to create a repeat dataset test bed for the evaluation of current and new software for the ability to consistently measure change in the volume of tumor-related T2/Fluid Attenuated Inversion Recovery (FLAIR) abnormality.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peters, M.D.; Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health Clinical Trials — https://www.dukehealth.org/clinical-trials